CLINICAL TRIAL: NCT02391714
Title: Nitrous Oxide for Pain Management of Intrauterine Device Insertion
Brief Title: Nitrous Oxide for Pain Management of Intrauterine Device (IUD) Insertion
Acronym: NIUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UNMHSC 13-289
Record Dates: First submitted 2015-03-05; First posted 2015-03-18 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Contraception
Keywords: pain assessment; patient satisfaction; Visual Analog Scale; contraceptive devices; nulliparity
MeSH Terms: conditions — Patient Satisfaction | interventions — Povidone-Iodine; Chlorhexidine; Oxygen; Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxygen (Placebo) (Placebo Comparator): 100% oxygen will be administered via disposable scented nasal masks 2 minutes before, throughout and 3-5 minutes after procedure.
  If you are randomized to this group, you will undergo the IUD insertion (including Povidone-Iodine or Chlorhexidine swab) using standard technique.
  Interventions: Procedure: IUD insertion; Drug: Povidone-Iodine; Drug: Chlorhexidine; Other: Oxygen
- Nitrous Oxide (NO) (Experimental): Nitrous Oxide in a fixed dose ratio of 50% nitrous/50% oxygen will be administered via disposable scented nasal masks 2 minutes before and throughout the procedure; 100% oxygen will be given after the procedure for 3-5 minutes.
  If you are randomized to this group, you will undergo the IUD insertion (including Povidone-Iodine or Chlorhexidine swab) using standard technique.
  Interventions: Procedure: IUD insertion; Drug: Povidone-Iodine; Drug: Chlorhexidine; Other: Nitrous oxide

INTERVENTIONS:
Procedure: IUD insertion — The IUD (Mirena® or ParaGard®) insertion procedure will occur in the usual manner for both arms. A bimanual exam will be performed, the speculum placed and the cervix visualized. The cervix will then by cleaned with iodine solution. If you are allergic to iodine, we will use chlorhexidine instead. A tenaculum will be placed on the cervix and a uterine sound will be used to measure cavity length. The Mirena® or ParaGard® IUD will be inserted with the specific introducer.
  Other Names: Mirena® insertion; ParaGard® insertion
Drug: Povidone-Iodine — Povidone-Iodine 10% w/w antiseptic swab for the cervix prior to IUD insertion.
  Other Names: PDI®
Drug: Chlorhexidine — For patients with allergy to iodine - 2% w/v chlorhexidine gluconate and 70% v/v isopropyl alcohol antiseptic swab for the cervix prior to IUD insertion.
  Other Names: ChloraPrep®
Other: Oxygen — 100% oxygen via nasal mask.
  Arms: Oxygen (Placebo)
Other: Nitrous oxide — Given in a fixed dose ratio of 50% nitrous oxide/50% oxygen via nasal mask.
  Arms: Nitrous Oxide (NO)

SUMMARY:
The purpose of this study is to determine whether Nitrous Oxide is effective in achieving pain control and satisfaction among nulliparous women getting the intrauterine device (IUD).

DETAILED DESCRIPTION:
Long acting reversible contraception (LARC) including the IUD provides several advantages that may be attractive to women. These include non-daily use, rapid reversibility and low failure rates. The American College of Obstetricians and Gynecologists (ACOG) endorses the use of IUDs among adolescents and nulliparous women, dispelling the myth that IUD use is contraindicated in this population.

Rates of IUD uptake among nulliparous women have not been reported. There are some barriers that may help explain the low uptake of IUDs by teens and nulliparous women, including fear of pain during IUD insertion. This concern is also voiced by providers who perceive pain with IUD insertion to be higher among nulliparous women (Allen, Goldberg et al. 2009).

There is limited evidence comparing subjective pain scores with IUD insertion between nulliparous versus parous women. However, there have been a number of studies evaluating the efficacy of misoprostol, non steroidal anti-inflammatory drugs and local anesthesia in reducing pain during IUD insertion. These included comparisons of pain scores between both nulliparous and multiparous women and reported pain scores by group. These studies have failed to demonstrate evidence that any of the aforementioned interventions significantly reduce pain scores compared to placebo (Allen et al. 2009). We conclude that pain with IUD insertion among nulliparous and adolescent women is within the high range of pain scale measurement standards. Therefore, further investigations of optimizing pain management during this procedure are warranted in order to lead to increased acceptability and adoption of IUDs among this population of women.

Nitrous oxide (NO) is an inhaled gas administered with oxygen in a fixed ratio for analgesia and sedation. It has been used for many years for procedural analgesia and anesthesia in outpatient settings and it reduces anxiety, the perception of pain and alters consciousness. It is attractive for the clinic setting as it demonstrates rapid induction and rapid resolution, allows for patient control of use, exhibits few side effects and boasts a benign safety profile in the setting of scavenging systems and open air clinics. Furthermore, NO systems are relatively inexpensive and noninvasive.

For all these reasons, NO seems to be an ideal approach for pain management with IUD insertion for nulliparous women. No studies have investigated the use of NO in this context. The aim of our study is to objectively identify pain reduction scores and satisfaction with NO use compared to typical insertion practices during IUD insertion for nulliparous women.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 OR between the ages of 12-17 with a parent/legal guardian who can consent
* English speaking
* Desires a Mirena® or ParaGard® IUD
* Nulliparous woman
* Can use laughing gas
* Has not taken narcotic pain medications prior to procedure

Exclusion Criteria:

* Currently pregnant
* If you have been pregnant before, pregnancy lasting longer than 19 weeks, 6 days
* Less than 4 weeks have elapsed from the end of a spontaneous abortion or medical abortion.
* Desires Skyla® IUD
* Pelvic Inflammatory Disease in the last 3 months
* Current mucopurulent discharge
* Uterine anomaly that distorts the uterine cavity
* Known uterine fibroid with disruption of the uterine cavity
* Copper allergy/Wilson's disease (for ParaGard®)
* Current cervical or uterine cancer
* Inability to breathe through the nose
* Significant active upper airway infection

Min Age: 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rameet Singh, MD MPH, Principal Investigator — UNM Division of Family Planning
Locations (1):
- Center for Reproductive Health, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Allen RH, Goldberg AB, Grimes DA. Expanding access to intrauterine contraception. Am J Obstet Gynecol. 2009 Nov;201(5):456.e1-5. doi: 10.1016/j.ajog.2009.04.027. Epub 2009 Jun 13. PMID 19527902
- [Background] Allen RH, Bartz D, Grimes DA, Hubacher D, O'Brien P. Interventions for pain with intrauterine device insertion. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD007373. doi: 10.1002/14651858.CD007373.pub2. PMID 19588429
- [Derived] Singh RH, Thaxton L, Carr S, Leeman L, Schneider E, Espey E. A randomized controlled trial of nitrous oxide for intrauterine device insertion in nulliparous women. Int J Gynaecol Obstet. 2016 Nov;135(2):145-148. doi: 10.1016/j.ijgo.2016.04.014. Epub 2016 Jul 16. PMID 27481016

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxygen (Placebo): 100% oxygen will be administered via disposable scented nasal masks 2 minutes before, throughout and 3-5 minutes after procedure.
  If you are randomized to this group, you will undergo the IUD insertion (including Povidone-Iodine or Chlorhexidine swab) using standard technique.
  IUD insertion: The IUD (Mirena® or ParaGard®) insertion procedure will occur in the usual manner for both arms. A bimanual exam will be performed, the speculum placed and the cervix visualized. The cervix will then by cleaned with iodine solution. If you are allergic to iodine, we will use chlorhexidine instead. A tenaculum will be placed on the cervix and a uterine sound will be used to measure cavity length. The Mirena® or ParaGard® IUD will be inserted with the specific introducer.
  Oxygen: 100% oxygen via nasal mask.
- Nitrous Oxide (NO): Nitrous Oxide in a fixed dose ratio of 50% nitrous/50% oxygen will be administered via disposable scented nasal masks 2 minutes before and throughout the procedure; 100% oxygen will be given after the procedure for 3-5 minutes.
  If you are randomized to this group, you will undergo the IUD insertion (including Povidone-Iodine or Chlorhexidine swab) using standard technique.
  IUD insertion: The IUD (Mirena® or ParaGard®) insertion procedure will occur in the usual manner for both arms. A bimanual exam will be performed, the speculum placed and the cervix visualized. The cervix will then by cleaned with iodine solution. If you are allergic to iodine, we will use chlorhexidine instead. A tenaculum will be placed on the cervix and a uterine sound will be used to measure cavity length. The Mirena® or ParaGard® IUD will be inserted with the specific introducer.
  Nitrous oxide: Given in a fixed dose ratio of 50% nitrous oxide/50% oxygen via nasal mask.
Period: Overall Study
Arm/Group | Oxygen (Placebo) | Nitrous Oxide (NO)
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxygen (Placebo) | Nitrous Oxide (NO) | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Full Range); unit: years] | 26.3 [17 to 40] | 24.93 [13 to 41] | 25.62 [13 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Mean Maximum Procedural Pain Scores
Description: Pain is assessed using a 0-100mm VAS with anchors 0 equals no pain and 100 equals worst pain imaginable. The minimal clinically important difference in pain for this study was set at 15mm.
Time Frame: 2 minutes after the procedure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxygen (Placebo) | Nitrous Oxide (NO)
Number analyzed (Participants) | 40 | 40
units on a scale | 55.3 (20.9) | 54.3 (24.8)

2. Secondary Outcome: Patient Satisfaction With Over-all Pain Control With IUD Insertion - VAS
Description: Satisfaction will be measured using a 100mm Visual Analog Scale (VAS), with anchors 0mm for very satisfied and 100mm for very dissatisfied.
Time Frame: Prior to clinic discharge, which is an average of 15 minutes after the procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Oxygen (Placebo): 100% oxygen will be administered via disposable scented nasal masks 2 minutes before, throughout and 3-5 minutes after procedure.
  If you are randomized to this group, you will undergo the IUD insertion (including Povidone-Iodine or Chlorhexidine swab) using standard technique.
  IUD insertion: The IUD (Mirena® or ParaGard®) insertion procedure will occur in the usual manner for both arms. A bimanual exam will be performed, the speculum placed and the cervix visualized. The cervix will then by cleaned with iodine solution. If you are allergic to iodine, we will use chlorhexidine instead. A tenaculum will be placed on the cervix and a uterine sound will be used to measure cavity length. The Mirena® or ParaGard® IUD will be inserted with the specific introducer.
  Povidone-Iodine: Povidone-Iodine 10% w/w antiseptic swab for the cervix prior to IUD insertion.
  Chlorhexidine: For patients with allergy to iodine - 2% w/v chlorhexidine gluconate and 70% v/v isopropyl alcohol antiseptic
- Nitrous Oxide (NO): Nitrous Oxide in a fixed dose ratio of 50% nitrous/50% oxygen will be administered via disposable scented nasal masks 2 minutes before and throughout the procedure; 100% oxygen will be given after the procedure for 3-5 minutes.
  If you are randomized to this group, you will undergo the IUD insertion (including Povidone-Iodine or Chlorhexidine swab) using standard technique.
  IUD insertion: The IUD (Mirena® or ParaGard®) insertion procedure will occur in the usual manner for both arms. A bimanual exam will be performed, the speculum placed and the cervix visualized. The cervix will then by cleaned with iodine solution. If you are allergic to iodine, we will use chlorhexidine instead. A tenaculum will be placed on the cervix and a uterine sound will be used to measure cavity length. The Mirena® or ParaGard® IUD will be inserted with the specific introducer.
  Povidone-Iodine: Povidone-Iodine 10% w/w antiseptic swab for the cervix prior to IUD insertion.
  Chlorhexidine: For patients
Arm/Group | Oxygen (Placebo) | Nitrous Oxide (NO)
Number analyzed (Participants) | 40 | 40
units on a scale | 60.3 (26.6) | 66.0 (32.2)

3. Secondary Outcome: Baseline Mean Pain Scores
Description: Baseline pain scores prior to IUD insertion is assessed using a 0-100mm VAS with anchors 0 equals no pain and 100 equals worst pain imaginable. The minimal clinically important difference in pain for this study was set at 15mm.
Time Frame: Before the IUD insertion procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxygen (Placebo) | Nitrous Oxide (NO)
Number analyzed (Participants) | 40 | 40
units on a scale | 1.9 (4.6) | 2.4 (4.1)

ADVERSE EVENTS:
Arm/Group | Oxygen (Placebo) | Nitrous Oxide (NO)
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No